CLINICAL TRIAL: NCT05411588
Title: A PHASE 1, RANDOMIZED, DOUBLE-BLIND, SPONSOR OPEN, PLACEBO-CONTROLLED, DOSE ESCALATING STUDY TO EVALUATE THE SAFETY, TOLERABILITY, PHARMACOKINETICS, AND PHARMACODYNAMICS OF SINGLE AND MULTIPLE INTRAVENOUS AND SUBCUTANEOUS DOSES OF PF-07275315 IN HEALTHY PARTICIPANTS
Brief Title: A Study to Learn How the Study Medicine Called PF-07275315 Works in Healthy People
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: C4531001; 2022-000854-27 (EudraCT Number)
Record Dates: First submitted 2022-06-06; First posted 2022-06-09 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Healthy Volunteers
Keywords: PF-07275315

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active (Experimental): PF-07275315
  Interventions: Drug: PF-07275315
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PF-07275315 — Active drug
  Other Names: No other name
  Arms: Active
Drug: Placebo — Placebo
  Other Names: No other name
  Arms: Placebo

SUMMARY:
The purpose of this clinical trial is to learn about the safety and effects of the study medicine (called PF-07275315) in healthy participants.

This study is seeking participants who:

* Are healthy as determined by medical evaluation.
* Are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Have a body mass index (BMI) of 17.5 to 32 kilogram per meter square - a total body weight of more than 50 kilograms (110 pounds)

Participants will be divided randomly into 8 different groups. All participants will receive either one PF-07275315 or a harmless treatment that has no medical effect (placebo) intravenous (IV) infusion (given directly into a vein). Participants will take part in this study for up to 541 days. During this time, eligible participants will receive single increasing amounts of PF-07275315 or placebo. Increase will only occur if the sponsor agrees that the next dose is likely to have acceptable safety and tolerability. The follow-up visit will take place 271 days after first treatment.

DETAILED DESCRIPTION:
This is an first-in-human within-cohort randomized, participant- and investigator-blind, sponsor-open, placebo-controlled study of the safety, tolerability, PK, and PD following single and multiple escalating doses of PF-07275315 that will be conducted in healthy adults.

ELIGIBILITY:
This study is seeking participants who:

* Are overtly healthy as determined by medical evaluation.
* Are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Have a body mass index (BMI) of 17.5 to 32 kg/m2; and a total body weight >50 kg (110 lb).

This study is not seeking participants who have:

* Evidence of active, latent, or inadequately treated infection with Mycobacterium tuberculosis (TB) as defined by both of the following
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C;
* Any of the following acute or chronic infections or infection history
* Any malignancies or have a history of malignancies with the exception of adequately treated or excised non-metastatic basal cell or squamous cell cancer of the skin, or cervical carcinoma in situ.
* Have undergone significant trauma or major surgery within 1 month of the first dose of study drug.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2022-06-09 (Actual); Primary Completion 2024-05-13 (Actual); Study Completion 2024-05-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with Adverse Events (AEs) | Baseline through study completion, approximately 561 days
  Incidence and severity of AEs
Number of participants with clinically meaningful change from baseline in laboratory Tests Results | Baseline through study completion, approximately 561 days
  Number of Participants With Change From Baseline in Laboratory Tests Results
Number of participants with clinically meaningful change from baseline in vital signs | Baseline through study completion, approximately 561 days
  Number of participants with change from baseline in vital signs
Number of participants with Serious AEs (SAEs) | Baseline through study completion, approximately 561 days
  Incidence and severity of SAEs
Number of participants with clinically meaningful change from baseline in ECG parameters | Baseline through study completion, approximately 561 days
  number of participants with change from baseline in ECG parameters

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | 1- 561 Days
  Cmax will be observed directly from data.
Time to Maximum Plasma Concentration (Tmax) of PF-07275315 | 1 - 561 Days
  Tmax will be observed directly from data.
Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUClast) of PF-07275315 | 1 - 561 Days
  Area under the plasma concentration-time curve from time 0 to the time of the last quantifiable concentration (AUClast)
Incidence of the development of Antidrug antibodies (ADA) against PF-07275315 | 1 - 561 Days
  To evaluate the immunogenicity profile of PF-07275315 in healthy adults.
Half-life of PF-07275315 | 1-561 days
  terminal elimination half-life will be measured
Area under the curve (AUC) of PF-07275315 serum concentration time-profile from time zero extrapolated to infinite time | 1-561 days
  AUCinf
AUC of PF-07275315 serum concentration time-profile over the dosing interval of 2 weeks or 336 hours | 1-561 days
  AUC336
Incidence of the development of neutralizing antibodies (NAb) against PF-07275315 | 1-561 days
  To evaluate the immunogenicity profile of PF-07275315 in healthy adults.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (4):
  - Orange County Research Center, Lake Forest, California
  - Orange County Research Center, Tustin, California
  - New Haven Clinical Research Unit, New Haven, Connecticut
  - Qps-Mra, Llc, South Miami, Florida
- Pfizer Clinical Research Unit - Brussels, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4531001